CLINICAL TRIAL: NCT01013311
Title: Efficacy if Implantable Cardioverter Defibrillators for the Prevention of Sudden Death in Patients With Cardiac Sarcoidosis
Brief Title: Implantable Cardiac Defibrillators for the Prevention of Sudden Death in Patients With Cardiac Sarcoidosis
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Stanford University (Other); Icahn School of Medicine at Mount Sinai (Other); Weill Medical College of Cornell University (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: HM12076
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Sarcoidosis of the Heart; Cardiomyopathy
Keywords: Implantable Cardioverter-Defibrillator (ICD)- pre-existing
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Sarcoidosis: Patients with Cardiac Sarcoidosis who had an ICD implanted

SUMMARY:
The purpose of this study is to identify patients with cardiac sarcoidosis who may be at risk for sudden death.

DETAILED DESCRIPTION:
Sarcoidosis is an inflammatory disease that can effect many organ systems. Patients with sarcoidosis involving the heart are at risk of sudden death related to ventricular arrythmias. However, we currently do not have a clinical test which can predict sudden cardiac death in these patients. While implantable cardioverter defibrillators(ICDs) can prevent sudden cardiac death in high risk patients, we do not know which patients will benefit from implantation of these devices. This clinical problem is important because we would like to identify patients at risk for sudden death who will benefit from ICD implantation. Additionally, we would like to avoid the risks to patients and financial expenses of inserting ICDs in patients who will not benefit from them.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cardiac Sarcoidosis
* Previous Implantable Cardioverter Defibrillator (ICD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-center retrospective study. Up to 20 Elctrophysiologists at Academic Centers across North America
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
retrospective collection of demographic and clinical data on patients with cardiac sarcoidosis who had an ICD implanted to correlate clinical variables with ICD therapies for ventricular arrhythmias | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Ellenbogen, MD, Principal Investigator — Virginia Commonweath University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Result] Banba K, Kusano KF, Nakamura K, Morita H, Ogawa A, Ohtsuka F, Ogo KO, Nishii N, Watanabe A, Nagase S, Sakuragi S, Ohe T. Relationship between arrhythmogenesis and disease activity in cardiac sarcoidosis. Heart Rhythm. 2007 Oct;4(10):1292-9. doi: 10.1016/j.hrthm.2007.06.006. Epub 2007 Jun 16. PMID 17905334
- [Result] Aizer A, Stern EH, Gomes JA, Teirstein AS, Eckart RE, Mehta D. Usefulness of programmed ventricular stimulation in predicting future arrhythmic events in patients with cardiac sarcoidosis. Am J Cardiol. 2005 Jul 15;96(2):276-82. doi: 10.1016/j.amjcard.2005.03.059. PMID 16018857
- [Result] Kron J, Sauer W, Schuller J, Bogun F, Crawford T, Sarsam S, Rosenfeld L, Mitiku TY, Cooper JM, Mehta D, Greenspon AJ, Ortman M, Delurgio DB, Valadri R, Narasimhan C, Swapna N, Singh JP, Danik S, Markowitz SM, Almquist AK, Krahn AD, Wolfe LG, Feinstein S, Ellenbogen KA. Efficacy and safety of implantable cardiac defibrillators for treatment of ventricular arrhythmias in patients with cardiac sarcoidosis. Europace. 2013 Mar;15(3):347-54. doi: 10.1093/europace/eus316. Epub 2012 Sep 21. PMID 23002195